CLINICAL TRIAL: NCT00250952
Title: A Randomized, Evaluator-Blinded, Two Centre Study of the Safety and Effect of Volume on the Diffusion and Efficacy of BOTOX Cosmetic™ (Botulinum Toxin Type A) in the Treatment of Lateral Orbital Rhytides.
Brief Title: Study to Determine If the Volume Used to Dilute BOTOX Cosmetic™ for Injection Affects Its Overall Effect and Duration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carruthers Dermatology Centre (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CCR-001
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2005-11-09 (Estimated); Status verified 2005-11

CONDITIONS: Skin Wrinkling
Keywords: Clinical Practice Variations
MeSH Terms: interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botox Cosmetic™

SUMMARY:
It is thought that the amount of fluid used to dilute Botox for injection has an effect on the quality of the result and the duration of effect on the treatment of upper face rhytides, even though the dose remains the same.

The study was designed to test this thinking, using the crow's feet wrinkles as the treatment area.

DETAILED DESCRIPTION:
It is thought that the amount of fluid used to dilute Botox for injection has an effect on the quality of the result and the duration of effect on the treatment of upper face rhytides, even though the dose remains the same.

20 female subjects (10 per site), who fit the inclusion/exclusion criteria for study participation were injected with 5 units of Botox (one injection each side) into the crow's feet area. The injections were prepared with one side randomly receiving a five fold difference in volume for dilution.

Response to treatment was evaluated at 14 days, 30 days, 60 days and 90 days after the injection visit. Standardized photography was taken at each visit.

Analysis of the photographs of the lateral orbital (crow's feet rhytides) at maximum attempted contraction (maximum smile) was done by Canfield Scientific, Inc., using a specialized software program created to detect and measure changes.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients; at least 18 years of age
* Subjects of childbearing potential must have a negative urine pregnancy test result at the Baseline/Screening Visit and practice a reliable method of contraception throughout the study.
* Bilaterally symmetric moderate (score 2 on Allergan Photonumeric Guide for Crow's Feet) Lateral Orbital Rhytides at maximum smile

Exclusion Criteria:

* Subjects who are pregnant, are planning a pregnancy during the study period, have an infant they are breast feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Subjects with a history of injection to the lateral orbital area with botulinum toxin type A within one year of baseline visit.
* Subjects with a history of adverse reaction to botulinum toxin type A.
* Subjects with a diagnosis of Myasthenia Gravis, Eaton-Lambert syndrome, Amyotrophic Lateral Sclerosis, or any other disease which might interfere with neuromuscular transmission.
* Subjects with a history of facial nerve palsy.
* Subjects with profound atrophy or excessive weakness of muscles in the target areas for injections.
* Subjects with a systemic infection or an infection at the injection site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-02; Study Completion 2005-06

PRIMARY OUTCOMES:
Using the per visit photographs, the effect of Botox was measured separately for each treatment site (right and left crow's feet at maximum smile) for all visits.

SECONDARY OUTCOMES:
Using the per visit photographs, the remaining effect of Botox treatment was measured separately for each treatment site (right and left crow's feet at maximum smile) for the 30, 60, and 90 day follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: J. Alastair Carruthers, MD, Principal Investigator — Carruthers Dermatology Centre, Inc.; Jeffrey S Dover, MD, Principal Investigator — Skin Care Physicians of Chestnut Hill
Locations (2):
- Skin Care Physicians of Chestnut Hill, Chestnut Hill, Massachusetts, United States
- Carruthers Dermatology Centre, Inc., Vancouver, British Columbia, Canada